CLINICAL TRIAL: NCT06148870
Title: Comparison of Efficacy Between Two Myopia Control Lenses
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Essilor International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: WS10356
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Myopia
Keywords: Refractive errors; Eye diseases; Axial length; Myopia Control
MeSH Terms: conditions — Myopia; Refractive Errors; Eye Diseases

STUDY DESIGN:
Intervention Model Description: This is a one-year, mono-centre, randomized, double-masked, monocular cross-over Clinical Trial with the objective to test and compare the efficacy of the new lens design in slowing down the increase of axial length and controlling myopic progression. The subject starts by wearing Myopia Control Lens 1 (MCL1) in one eye, and Myopia Control Lens 2 (MCL2) in another eye. After 6 months, a new pair of study spectacles will be dispensed with MCL1 and MCL2 crossed over. At the end of the 1-year period, each eye would have worn both MCL1 and MCL2 for 6 months each. There will be a total of 7 study visits with follow up periods at 3 months, 6 months and 12 months
Who Masked: Participant, Investigator
Masking Description: As this is a double-masked, randomized controlled trial, both the investigators and subjects will be masked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MCL1 (Active Comparator): The MCL1 is a myopia control lens that will be worn in one eye for 6 months.
  Interventions: Device: Myopia Control Lens-1 (MCL1); Device: Myopia Control Lens-2 (MCL2)
- MCL2 (Experimental): The MCL2 is a myopia control lens that will be worn on the contralateral eye for 6 months.
  Interventions: Device: Myopia Control Lens-1 (MCL1); Device: Myopia Control Lens-2 (MCL2)

INTERVENTIONS:
Device: Myopia Control Lens-1 (MCL1) — The MCL1, is a myopia control lens that corrects refractive error and simultaneously creates myopia control signals. It will be worn on one eye for 6 months.
Device: Myopia Control Lens-2 (MCL2) — The MCL2, is a myopia control lens that corrects refractive error and simultaneously creates myopia control signals. It will be worn on the contralateral eye for 6 months.

SUMMARY:
This is a one-year, mono-centre, randomize, double-masked, monocular cross-over clinical trial designed to test and compare the efficacy of the new lens design in slowing down the increase of axial length and controlling myopia progression.

DETAILED DESCRIPTION:
The clinical trial aims to assess the safety and efficacy of a test lens, designed to modify the amount of myopic control signal on the retina without compromising vision. The primary goal of this clinical trial is to evaluate the effectiveness of the test lens in slowing down the increase of axial length and controlling myopia progression compared to the reference lens design.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer subject and guardian, fluent English spoken, willing to follow protocol and able to read, comprehend and sign the informed consent & assent form.
* Equal to or greater than 6 years and not older than 11 years at time of informed consent and assent.
* Spherical equivalent refractive error (SER) by manifest refraction between -0.50 and -4.75 D in each eye.
* Astigmatism, if present, of not more than 2.00 D.
* Difference in SER between the two eyes (Anisometropia) by manifest refraction not more than 1.00 D.
* Best corrected visual acuity in each eye better than +0.20 logMAR
* Agree to wear study spectacles for at least 10 hours a day and 6 days a week
* Willingness and ability to participate in trial for 1 year
* Willingness and ability to attend scheduled visits
* Not to involve concurrently in other myopia control treatments

Exclusion Criteria:

* History or presence of an Ocular disease, Strabismus, Amblyopia
* Undergoing any myopia control intervention specifically Atropine and Orthokeratology
* History of myopia control intervention specifically Atropine, Orthokeratology

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Change in Axial Length | 12 months
  To evaluate the effectiveness of the MCL2 in slowing myopia progression with respect to the change in Axial Length (AL) from baseline compared to MCL1 at 12-month.

SECONDARY OUTCOMES:
Change in Spherical Equivalent Refraction | 12 months
  To evaluate the effectiveness of the MCL2 lens in slowing myopia progression with respect to the change in Spherical Equivalent Refraction (SER) from baseline compared to MCL1 at 12-month.

CONTACTS AND LOCATIONS:
Overall Officials: Wee Sing Ong, Principal Investigator — Essilor R&D Centre Singapore
Locations (1):
- Essilor R&D Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holden BA, Fricke TR, Wilson DA, Jong M, Naidoo KS, Sankaridurg P, Wong TY, Naduvilath TJ, Resnikoff S. Global Prevalence of Myopia and High Myopia and Temporal Trends from 2000 through 2050. Ophthalmology. 2016 May;123(5):1036-42. doi: 10.1016/j.ophtha.2016.01.006. Epub 2016 Feb 11. PMID 26875007
- [Background] Bao J, Huang Y, Li X, Yang A, Zhou F, Wu J, Wang C, Li Y, Lim EW, Spiegel DP, Drobe B, Chen H. Spectacle Lenses With Aspherical Lenslets for Myopia Control vs Single-Vision Spectacle Lenses: A Randomized Clinical Trial. JAMA Ophthalmol. 2022 May 1;140(5):472-478. doi: 10.1001/jamaophthalmol.2022.0401. PMID 35357402
- [Background] Smith EL 3rd. Optical treatment strategies to slow myopia progression: effects of the visual extent of the optical treatment zone. Exp Eye Res. 2013 Sep;114:77-88. doi: 10.1016/j.exer.2012.11.019. Epub 2013 Jan 3. PMID 23290590